CLINICAL TRIAL: NCT01812655
Title: Comparison of Virtual Reality and Passive Distraction on Burn Wound Care
Brief Title: Comparison of Virtual Reality and Passive Distraction on Burn Wound Care Pain in Adolescents
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Early termination of study due to fewer subjects available than expected resulting in small sample size.
Sponsor: University of Arkansas (Other)
Collaborators: Arkansas Children's Hospital Research Institute (Other); Arkansas Biosciences Institute (Unknown); Arkansas Children's Hospital Burn Center (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 109422
Record Dates: First submitted 2013-03-13; First posted 2013-03-18 (Estimated); Results first posted 2013-08-06 (Estimated); Last update posted 2013-08-06 (Estimated); Status verified 2013-08

CONDITIONS: Burns; Wound Care; Pain
Keywords: pain; anxiety; children; adolescents; burn; virtual reality; distraction
MeSH Terms: conditions — Burns; Pain; Anxiety Disorders

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Virtual Reality (Experimental): Virtual reality using a software program designed for burn patients during burn wound care
  Interventions: Device: Virtual Reality
- Passive distraction (Active Comparator): watching a movie
  Interventions: Other: Passive Distraction
- UC provided by the nurses (No Intervention)

INTERVENTIONS:
Device: Virtual Reality
  Arms: Virtual Reality
Other: Passive Distraction
  Arms: Passive distraction

SUMMARY:
Relief of severe burn wound care pain may require both medications to relieve pain and non-medication interventions,such as distraction. Little is known about distraction's effectiveness. Virtual reality may be an effective distraction. The aims of this study are 1)to evaluate the effect of virtual reality (VR), a newer interactive kind of distraction, compared to passive distraction (PD) by watching a movie, and usual care (SC) that is provided by the nurses, on pain experienced by adolescents during burn wound care and 2)to determine the relationship among anxiety, desire for distraction, and engagement with distraction on the pain.

ELIGIBILITY:
Inclusion Criteria:

* undergoing burn wound care in the Arkansas Children's Hospital (ACH) outpatient burn clinic;
* first time visit to the ACH outpatient burn clinic or first clinic visit without conscious sedation;
* adolescents ages 10 to 17 years;
* English speaking;
* absence of a history of motion sickness (motion sickness has been reported in some VR users);
* absence of a seizure disorder (because prolonged immersion in VR may lead to seizures and vertigo in individuals with seizure disorders, these individuals will be excluded from the study);
* absence of a cognitive developmental disability determined on prescreening by presence of a Section 504 accommodation plan or Title VIII individualized educational plan (IEP) in school. If the parent identifies the nature of the IEP or 504 plan as unrelated to a cognitive delay, then the child or adolescent will be included in the study.

Exclusion Criteria:

* Burns that would interfere with study procedures
* Incarcerated minors
* Children in foster care

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra A Jeffs, PhD, RN, Principal Investigator — Arkansas Children's Hospital Research Institute
Locations (1):
- Arkansas Children's Hospital, Little Rock, Arkansas, United States

REFERENCES:
- [Background] Askay SW, Patterson DR. What are the psychiatric sequelae of burn pain? Curr Pain Headache Rep. 2008;12(2):94-97. Das DA, Grimmer KA, Sparnon AL, et al. The efficacy of playing a virtual reality game in modulating pain for children with acute burn injuries: a randomized controlled trial. BMC Pediatr. 2005;5(1):1471-2431. Patterson DR, Weichman SA, Jensen MP, et al. Hypnosis delivered through immersive virtual reality for burn pain: a clinical case series. Int J Clin Exp Hypn. 2006;54(2):130-142. Hoffman HG, Chambers GT, Meyer WJ, et al. Virtual reality as an adjunctive non-pharmacologic analgesic for acute burn pain during medical procedures. Ann. Behav. Med. 2011;41(2):183-191. doi: 10.1007/s12160-010-9248-7. Smith JS, Smith KR, Rainey SL. The psychology of burn care. J Trauma Nurs. 2006;13(3):105-106.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited from 6/2010 until 4/2012 in the outpatient Burn Center clinic.
Pre-assignment Details: One participant was re-assigned to standard care prior to group assignment when the virtual reality (VR) equipment failed during set-up.
Groups:
- Virtual Reality: Patients were distracted from their burn wound care pain throughout their entire burn wound care procedure using an interactive virtual reality program designed for burn patients. Mean time for the intervention was 31.6 minutes.
- Passive Distraction: Patients watched a movie, Cloudy with a Chance of Meatballs, throughout their burn wound care to offer passive distraction from wound care pain. Mean time for the intervention use was 31.6 minutes.
- SC Provided by the Nurses: Nurses provided their usual, standard care throughout the entire burn wound care, such as talking with the patients. Mean time for the intervention use was 49.0 minutes.
Period: Overall Study
Arm/Group | Virtual Reality | Passive Distraction | SC Provided by the Nurses
Started | 9 (Virtual Reality-Patients used an interactive VR program during their burn wound care procedure.) | 11 (Passive Distraction-Patients watched a movie during their burn wound care.) | 10 (Nurses provided their usual, standard care throughout the entire burn wound care.)
Completed | 8 | 10 | 10
Not Completed | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Virtual Reality | Passive Distraction | Standard Care Provided by the Nurses | Total
Number analyzed (Participants) | 9 | 11 | 10 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 9 | 11 | 10 | 30
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 14.3 (2.0) | 12.6 (2.1) | 13.9 (2.8) | 13.5 (2.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 2 | 2 | 9
  Male | 4 | 9 | 8 | 21
Region of Enrollment [Number; unit: participants]
  United States | 9 | 11 | 10 | 30
STAIC - State Anxiety [Mean (Standard Deviation); unit: Scores on a scale] — Participants self-rated 20 statements about how the individual feels at the present moment with responses provided on a three-point rating scale. Total scores on the scale range from 20-60.
  Scores on a scale | 34.4 (9.1) | 27.0 (4.0) | 33.6 (10.6) | 31.5 (8.7)
STAIC - Trait Anxiety [Mean (Standard Deviation); unit: Scores on a scale] — Participants self-rated 20 statements on a three-point rating scale that best described how the person usually feels. Total scores on the scale range from 20-60.
  Scores on a scale | 34.6 (5.0) | 33.5 (7.5) | 34.1 (7.1) | 34.0 (6.5)
Pre-Procedure Pain [Mean (Standard Deviation); unit: Score on a scale] — Participants rated pre-procedure pain on the Adolescent Pediatric Pain Tool word graphic rating scale with no pain and worst possible pain as anchors on the 0-100mm scale.
  Score on a scale | 40.1 (30.9) | 8.7 (14.5) | 22.9 (26.0) | 22.8 (26.6)

OUTCOME MEASURES:

1. Primary Outcome: Self-reported Wound Care Procedure Pain Score
Description: The acute pain experienced during the burn wound care procedure was measured on a 100mm visual analog scale called the Adolescent Pediatric Pain Tool through self-report by adolescents ages 10-17 years receiving outpatient burn wound care. The scale ranges from 0mm (No Pain) to 100mm (Worst Pain).
Time Frame: Within the first 20 minutes following completion of the burn wound care procedure
Population: Intention to treat
Measure: Least Squares Mean (95% Confidence Interval); unit: mm
Arm/Group | Virtual Reality | Passive Distraction | Standard Care Provided by the Nurses
Number analyzed (Participants) | 8 | 10 | 10
mm | 28.7 [14.1 to 43.3] | 52.4 [40.3 to 64.5] | 38.4 [27.4 to 49.4]
Statistical Analysis 1: Comparison: Virtual Reality vs Passive Distraction; Test type: Superiority or Other; p = 0.029, Regression, Linear; Mean Difference (Final Values) = 23.7, 95% CI 2-sided [2.4 to 45.0] — Mean difference = PD group - VR group
Statistical Analysis 2: Comparison: Virtual Reality vs Standard Care Provided by the Nurses; Test type: Superiority or Other; p = 0.32, Regression, Linear; Mean Difference (Final Values) = 9.7, 95% CI 2-sided [-9.5 to 28.9] — Mean difference = VR group - SC group

2. Secondary Outcome: Desire for Distraction
Description: Participants were asked "I wanted to be distracted from during my treatment today." (Agree-Disagree) from the Post-Procedure Questionnaire
Time Frame: Post-procedure (approximately 30-75 minutes)
Measure: Number; unit: participants
Arm/Group | Virtual Reality | Passive Distraction | SC Provided by the Nurses
Number analyzed (Participants) | 8 | 10 | 10
participants
  Yes | 7 | 7 | 7
  No | 0 | 2 | 3
  Did not Answer Question | 1 | 1 | 0
Statistical Analysis 1: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = .26, Semipartial correlation; Semipartial correlation = 0.223 — Semipartial correlation between desire for distraction and STAIC State Anxiety measured at Baseline for all participants
Statistical Analysis 2: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = .59, Semipartial correlation; Semipartial correlation = 0.119 — Semipartial correlation between desire for distraction and STAIC Trait Anxiety measured at Baseline for all participants
Statistical Analysis 3: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = .60, Semipartial correlation; Semipartial correlation = -0.059 — Semipartial correlation between desire for distraction and Procedural Pain (Outcome Measure #1) for all participants

3. Secondary Outcome: Engagement With Distraction and Belief in Distraction's Efficacy
Description: For Engagement with Distraction,VR and PD participants were asked on the Post-testing Questionnaire: "Were you able to pay attention to the DVD or to the VR during your burn treatment?" (1=could not pay attention at all; 5=totally absorbed at all times)
  For Belief in Distraction's Efficacy, VR and PD participants were asked on the Post-Procedure Questionnaire: "I believe that the distraction lessened my pain during my burn treatment today." (on a scale of 1=Distraction did not help to lessen my pain at all; 5=Distraction completely helped to lessen my pain at all times)
Time Frame: Post-procedure (approximately 30-75 minutes)
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Virtual Reality | Passive Distraction | SC Provided by the Nurses
Number analyzed (Participants) | 8 | 10 | 10
scores on a scale
  Engagement with Distraction | 3.6 (0.9) | 2.6 (1.1) | NA (NA) — Participants were not asked because not applicable.
  Belief in Distraction's Efficacy | 2.9 (1.2) | 2.6 (1.0) | NA (NA) — Participants were not asked because not applicable.
Statistical Analysis 1: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = 0.15, Semipartial Correlation; semipartial correlation = -0.276 — Semipartial correlation between Engagement with Distraction and STAIC State Anxiety measured at Baseline for all participants
Statistical Analysis 2: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = 0.18, Semipartial correlation; Semipartial correlation = -0.347 — Semipartial correlation between Engagement with Distraction and STAIC Trait Anxiety measured at Baseline for all participants
Statistical Analysis 3: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = 0.054, Semipartial correlation; Semipartial correlation = 0.210 — Semipartial correlation between Engagement with Distraction and Procedural Pain (Outcome Measure #1) for all participants
Statistical Analysis 4: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = 0.61, Semipartial Correlation; Semipartial Correlation = -0.102 — Semipartial correlation between Belief in Distraction's Efficacy and STAIC State Anxiety measured at Baseline for all participants
Statistical Analysis 5: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = 0.007, Semipartial Correlation; Semipartial Correlation = -0.622 — Semipartial correlation between Belief in Distraction's Efficacy and STAIC Trait Anxiety measured at Baseline for all participants
Statistical Analysis 6: Comparison: Virtual Reality vs Passive Distraction vs SC Provided by the Nurses; Test type: Superiority or Other; p = 0.045, Semipartial correlation; Semipartial correlation = -0.217 — Semipartial correlation between Belief in Distraction's Efficacy and Procedural Pain (Outcome Measure #1) for all participants

ADVERSE EVENTS:
Arm/Group | Virtual Reality | Passive Distraction | UC Provided by the Nurses
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Early termination of study due to fewer subjects available than expected resulting in small sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No